CLINICAL TRIAL: NCT00945373
Title: Combination Therapy for the Treatment of Erythematotelangiectatic Rosacea
Brief Title: Combination Therapy for the Treatment of Rosacea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ellen Marmur (Other)
Collaborators: American Society for Laser Surgery and Medicine (Other)
Responsible Party: Sponsor-Investigator, Ellen Marmur, Principal Investigator, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO # 09-0839
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Erythematotelangiectatic Rosacea
Keywords: rosacea; telangiectasias; topical treatment; pulsed dye laser
MeSH Terms: conditions — Rosacea; Telangiectasis | interventions — Calcium Dobesilate; Lasers, Dye

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erythematotelangiectatic Rosacea (Experimental): 2.5% gel calcium dobesilate and pulsed dye laser
  Interventions: Drug: calcium dobesilate; Procedure: pulsed dye laser

INTERVENTIONS:
Drug: calcium dobesilate — 2.5% gel
Procedure: pulsed dye laser — All study patients will be treated with 595 nm PDL (Vbeam, Candela Corp, Wayland, Mass) with an initial test spot using a fluence of 10 J/cm2, 7-mm spot size and 1.5-ms pulse duration. Based on the biologic response of the test area, the fluence will accordingly be adjusted up or down to find a fluence that produces a transient purpuric effect for a few seconds only.

SUMMARY:
The purpose of this study is to determine the efficacy of calcium dobesilate in combination with pulsed dye laser for the treatment of rosacea.

DETAILED DESCRIPTION:
Rosacea is a common cutaneous disorder characterized by facial erythema, papules and pustules and telangiectasias. The clinical manifestations of this disorder are distributed along the convexities of the face such as the cheeks, chin, nose and central aspects of the forehead.

The flushing and telangiectasias associated with erythematotelangietatic rosacea (ETR) are notoriously difficult to treat with standard medications. Patients with ETR have a lower threshold for irritation from topically applied drugs and these substances may even exacerbate their symptoms.

Pulsed dye laser (PDL) is widely considered as the treatment of choice for vascular malformations including telangiectasias, port wine stains and hemangiomas. Several studies have shown successful treatment of rosacea-associated telangiectasia and erythema with pulsed dye laser. Moreover, calcium dobesilate (2,5-dihydroxybenzene sulfonate) is a drug that inhibits vascular smooth muscle cell growth and inhibits cellular proliferation. As a synthetic inhibitor of fibroblast growth factor (FGF), calcium dobesilate targets angiogenic growth factors which lead to uncontrolled blood vessel growth. In light of the fact that angiogenesis has been implicated in erythematotelangietatic rosacea, calcium dobesilate will be useful in the treatment of this subtype of rosacea.

Thus, combination treatment with PDL and calcium dobsilate will act in a synergistic manner to reduce the erythema, flushing and telangectasia associated with erythematotelangietatic rosacea.

If the subject meets the inclusion criteria and informed consent is obtained, the subject will receive 2.5% calcium dobesilate get to apply to half of the face (randomized). The subject will also receive pulsed dye laser treatments to the whole face at two week intervals for a maximum of 3 treatments. The primary endpoint of this study will be the severity of rosacea at the end of the 20 week study.

ELIGIBILITY:
Inclusion Criteria:

1. Must understand and voluntarily sign an informed consent form.
2. Must be male or female and aged ≥ 18 years at time of consent.
3. Must be able to adhere to the study visit schedule and other protocol requirements.
4. Must have clinically typical confirmed diagnosis of erythematotelangestatic rosacea.
5. Females of childbearing potential (FCBP)‡ must have one negative urine pregnancy tests at screening. In addition, sexually active FCBP must agree to use TWO of the following adequate forms of contraception while on study medication: oral, injectable, or implantable hormonal contraceptives; tubal ligation; intrauterine device; barrier contraceptive with spermicide; or vasectomized partner while on the study. A FCBP must agree to have pregnancy tests every 4 weeks while on study medication.
6. Males (including those who have had a vasectomy) must agree to use barrier contraception (latex condoms) when engaging in sexual activity with FCBP while on study medication.

Exclusion Criteria:

1. Inability to provide voluntary informed consent.
2. Pregnant or breastfeeding female.
3. A skin examination reveals the presence of another skin disease and/or condition (excessive facial hair, excessive scarring, sunburn, or other disfigurement) located on the face that would confound the evaluation of the rosacea.
4. Current or past ocular rosacea, such as conjunctivitis, iritis and keratitis of sufficient severity to require topical or systemic antibiotics.
5. Subjects with recurrent gastritis, renal dysfunction or ulcer disease (peptic or duodenal).
6. Treatment with topical antibiotics, topical steroids, topical retinoids and other topical rosacea treatments on the face within 14 days of baseline and throughout the study.
7. Treatment with any systemic medication or therapy known to affect inflammatory responses within the 30 days prior to baseline and throughout the study.
8. Treatment with systemic retinoids within 6 months prior to study entry (e.g., acitretin, isotretinoin).
9. Use of laser or light based rosacea treatments within the past 2 months.
10. History of hypersensitivity or allergies to any ingredient in the study drug.
11. Current drug or alcohol abuse.
12. Have participated in any clinical trial involving an investigational drug or cosmetic product or procedure within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-07; Primary Completion 2010-05 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Investigator Global Assessment (IGA) scale | one year
  Global rosacea scale assssed as the success of rosacea treatment is usually defined as a score of 1 ('almost clear') or 0 ('clear') on the 5-point Investigator Global Assessment (IGA) scale. full scale from 0-4, with higher score indicating more disease.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Marmur, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States